CLINICAL TRIAL: NCT07297069
Title: Combination of INFLIXIMAB With TOFACITINIB in ASUC - CINTO Trial
Brief Title: Combination Therapy With Infliximab and Tofacitinib for Acute Severe Ulcerative Colitis - CINTO Trial
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Mohan Ramchandani, Senior Registrar, Asian Institute of Gastroenterology, India
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CINTO 1
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Acute Severe Ulcerative Colitis
Keywords: Rescue therapy; Combination therapy; Steroid refractory ulcerative colitis; Infliximab; Tofacitinib
MeSH Terms: interventions — Infliximab; tofacitinib

STUDY DESIGN:
Intervention Model Description: Three arm parallel randomized pilot trial comparing infliximab alone, tofacitinib alone, and combination therapy with infliximab plus tofacitinib in adults hospitalized with acute severe ulcerative colitis who do not respond to intravenous corticosteroids.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Infliximab Plus Tofacitinib (Experimental): Participants with acute severe ulcerative colitis who do not respond to intravenous corticosteroids will receive combination therapy with infliximab and tofacitinib. Infliximab 300 mg will be given intravenously, and tofacitinib will be administered orally at 10 mg twice daily. This arm evaluates whether combination therapy produces enhanced early clinical improvement and offers greater effectiveness and safety in inducing early clinical remission and mucosal healing compared with either agent alone.
  Interventions: Drug: Infliximab; Drug: Tofacitinib
- Infliximab Only (Active Comparator): Participants with acute severe ulcerative colitis who do not respond to intravenous corticosteroids will receive infliximab alone as rescue therapy. Infliximab will be administered at a dose of 300 mg intravenously according to protocol. This arm evaluates the effectiveness and safety of infliximab monotherapy in inducing early clinical remission and mucosal healing.
  Interventions: Drug: Infliximab
- Tofacitinib Only (Active Comparator): Participants with acute severe ulcerative colitis who do not respond to intravenous corticosteroids will receive tofacitinib alone as rescue therapy. Tofacitinib will be administered orally at 10 mg twice daily. This arm assesses the effectiveness and safety of tofacitinib monotherapy in inducing early clinical remission and mucosal healing.
  Interventions: Drug: Tofacitinib

INTERVENTIONS:
Drug: Infliximab — Participants with acute severe ulcerative colitis who do not respond to intravenous corticosteroids will receive infliximab as rescue therapy. Infliximab 300 mg will be administered intravenously. This arm evaluates the effectiveness and safety of infliximab monotherapy in inducing early clinical remission and mucosal healing.
  Arms: Infliximab Only; Infliximab Plus Tofacitinib
Drug: Tofacitinib — Participants with acute severe ulcerative colitis who do not respond to intravenous corticosteroids will receive tofacitinib as rescue therapy. Tofacitinib will be administered orally at 10 mg twice daily. This arm assesses the effectiveness and safety of tofacitinib monotherapy in inducing early clinical remission and mucosal healing.
  Arms: Infliximab Plus Tofacitinib; Tofacitinib Only

SUMMARY:
In adults hospitalized with acute severe ulcerative colitis who fail to respond to intravenous steroids, does treatment with a combination of infliximab and tofacitinib, compared with infliximab alone or tofacitinib alone, result in higher rates of early clinical remission and mucosal healing, and fewer treatment-related complications over a 10 week period

DETAILED DESCRIPTION:
Acute severe ulcerative colitis (ASUC) is a life threatening manifestation of ulcerative colitis that requires urgent medical treatment and hospitalization. Despite the use of rapid induction intravenous corticosteroids, some patients fail to respond and require rescue therapy. Infliximab is commonly used as rescue treatment; however, its effectiveness may be reduced in patients with severe inflammation and hypoalbuminemia. As a result, colectomy rates for ASUC remain significant and improved early rescue strategies are needed.

Tofacitinib is an oral Janus kinase inhibitor that targets multiple cytokine pathways involved in ulcerative colitis. It has a rapid onset of action and has shown benefit in severe and steroid-refractory disease. Because infliximab and tofacitinib act on different immunologic targets, their combined use may provide complementary therapeutic effects. Emerging observational data suggest that combining a biologic agent with a small-molecule therapy may be safe and potentially more effective in patients with severe disease who are at high risk for treatment failure.

This study is designed to explore whether the combination of infliximab and tofacitinib offers greater early clinical benefit compared to infliximab alone, tofacitinib alone for adults hospitalized with ASUC who do not respond to intravenous corticosteroids.The goal is to generate preliminary data that may inform future treatment approaches aimed at improving remission rates, accelerating mucosal healing, and reducing the need for colectomy in this high risk population.

ELIGIBILITY:
Inclusion Criteria:

Adult (aged 18 years to 65 years) patients hospitalised due to ASUC

Exclusion Criteria:

1. Patients with UC who did not meet the Truelove Witts criteria for ASUC.
2. Patients who are already on Tofacitinib / Infliximab.
3. Latent or active tuberculosis.
4. Crohn's or Indeterminate colitis.
5. Mega colon (if the diameter of the transverse colon is 5.5 cm or more, with apparent oedema of the bowel wall on plain abdominal radiographs).
6. Pseudomembranous colitis or concomitant CMV colitis.
7. Intestinal perforation.
8. Massive haemorrhage requiring emergency colectomy.
9. Pregnant or lactating female individuals.
10. Current diagnosis or history of thromboembolic disease patients with severe cardiorespiratory, renal or hepatic Co morbidities.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Remission Rate | Week 1 and Week 4
  Clinical remission is defined as defined as a Mayo score ≤2 and no individual subscore >1.Participants meeting these criteria will be classified as achieving clinical remission.

SECONDARY OUTCOMES:
Clinical Response Rate | Week 1 and Week 4
  Reduction of baseline Mayo score by ≥3 points and a decrease of 30% from the baseline score with a decrease of at least one point on the rectal bleeding subscale or an absolute rectal bleeding score of 0 or 1.
Mucosal Healing Rate | Week 4 and Week 12
  Mucosal healing is defined as an endoscopic Mayo score of 0 or 1 on flexible sigmoidoscopy. Participants undergoing endoscopic evaluation who meet these criteria will be classified as achieving mucosal healing.
Treatment Related Adverse Events | Baseline through Week 12
  Adverse events related to study medications, including but not limited to infections, lymphocytopenia, thromboembolic events, hyperlipidemia, and infusion or drug-related reactions, will be recorded throughout the study period. Severity and relationship to the study intervention will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Vamsi Krishna Ankam, DrNB(gastroenterology), Principal Investigator — Asian Institute of Gastroenterology, Hyderabad
Locations (1):
- Asian Institute of Gastroenterology, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because data sharing is not planned for this study.

REFERENCES:
- [Background] Hickman K, Jordan R, Sonnier W. Combination biologic and small molecule therapy for refractory ulcerative colitis. Gastroenterology. 2022;162(3 Suppl):S103.
- [Background] A genome-scale CRISPR tool for targeting multiple gene family members at once. Nat Plants. 2023 Apr;9(4):511-512. doi: 10.1038/s41477-023-01388-y. No abstract available. PMID 36973416